CLINICAL TRIAL: NCT05676983
Title: Investigation of the Effects of Balance Discs With Different Surfaces Used in Balance Education in Children With Cerebral Palsy
Brief Title: Investigation of the Effects of Balance Discs With Different Surfaces Used in Balance Education in Children With Cerebral Palsy on Proprioceptive Sense and Balance.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, İlkan Cicek, Postgraduate-physiotherapy graduate student, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PTIlkan
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiky balance disc study group (Experimental): Bobath therapy will be studied with the children in this group and balance training will be given on the rough (spiky) surface of the extra balance disc.
  Interventions: Other: Pediatric neurodevelopmental therapy; Other: smooth balance disc
- Smooth balance disc study group (Experimental): Bobath therapy will be studied with the children in this group and balance training will be given on the smooth (flat) surface of the extra balance disc.
  Interventions: Other: Spiky balance disc; Other: Pediatric neurodevelopmental therapy

INTERVENTIONS:
Other: Spiky balance disc — Balance discs consist of smooth and rough surface. Balance training is given to children with cerebral palsy on these two surfaces. Thanks to its balance disc structure, it plays an active role in the development of balance.
  Arms: Smooth balance disc study group
Other: Pediatric neurodevelopmental therapy — Bobath therapy
Other: smooth balance disc — Balance discs consist of smooth and rough surface. Balance training is given to children with cerebral palsy on these two surfaces. Thanks to its balance disc structure, it plays an active role in the development of balance.
  Arms: Spiky balance disc study group

SUMMARY:
This is a non-invasive prospective study investigating the effects of balance discs with different surfaces used in balance education in children with cerebral palsy on proprioceptive sense and balance.

DETAILED DESCRIPTION:
Many methods are used for balance training. One of them is balance discs. Balance discs consist of smooth and rough surfaces. Balance training is given to children with cerebral palsy on these two surfaces. Thanks to its balance disc structure, it plays an active role in the development of balance, but there is a need for evidence about whether rough or smooth surfaces and training have superiority over each other. Knowing the difference between the two surfaces will help the staff about which surface to use in the treatment and will be beneficial for the children.

The aim of this study is to determine whether there is a difference between a rough and smooth surface in terms of improving proprioceptive sense and balance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy
* Diagnosed with motor developmental delay
* 0-12 years old
* Levels 1 and 2 according to GMFCS
* Having bilateral and unilaterally affected spastic type CP
* Cooperate with assessments

Exclusion Criteria:

* Botulinum toxin administration in the last 6 months
* Having had any surgical operation in the last 6 months
* Having dyskinetic, ataxic and hypotonic type CP
* Unable to cooperate with assessments

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-01-09 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Berg balance test: | baseline and week 10
  The Pediatric Berg Balance Test is a modified version of the Berg Balance Test used to assess functional balance skills in school-aged children.Patients are evaluated out of 56 points, with the highest score being 56. Change will be evaluated
Change in Functional reach test | baseline and week 10
  The Functional Reach Test is a clinical outcome measurement and assessment tool to detect dynamic balance in a single simple task. While standing, it measures the distance between the length of an extended arm at maximum forward reach while maintaining a stable base of support.Change will be evaluated.
Change in One-leg standing test | baseline and week 10
  The one-leg stance test is a test in which the time to stand on balance is measured on the right and left extremities of the patient, and evaluates the static balance. Change will be evaluated.
Change in Proprioceptive sensory test: | baseline and week 10
  Active and passive repositioning test will be used to evaluate ankle proprioceptive sensation.
  Passive repositioning: The person to be tested is asked to learn that position by positioning the joint at a certain angle. Then, while the joint is moved passively, the person is asked to stop the movement when it reaches the previously learned position. The numerical difference between the angle found by the person and the angle taught before is evaluated.
  Active repositioning: The person is asked to find the position taught to the person by moving their extremity, and the numerical difference is determined.Change will be evaluated.

OTHER OUTCOMES:
height | baseline
  Children's height will be measured in cm with a tape measure.
weight | baseline
  Their weight will be measured with precision scales and indicated in kg.
body mass index | baseline
  Body mass index will be stated as kilo/meter*2.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal Üniversitesi, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bezgin S, Akkaya KU, Cicek I, Akbas Y, Elbasan B. Effects of balance training on different surfaces on ankle proprioception and functional balance in children with spastic cerebral palsy: a single-blind randomized controlled trial. BMC Pediatr. 2026 Jan 3;26(1):3. doi: 10.1186/s12887-025-06346-5. PMID 41485031